CLINICAL TRIAL: NCT07241299
Title: Understanding Chronic Treatments by Patients Over 65 Years of Age
Acronym: ordonnance
Status: Recruiting | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2025_RIPH_02_ordonnance
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Chronic Treatments
Keywords: chronic treatments; patients over 65 years
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — Data collection

SUMMARY:
The ageing of the French population is accompanied by an increase in the number of chronic conditions per person. In 2008, according to IRDES (Institute for Research and Documentation in Health Economics), the average number of reported illnesses was six for people over the age of 65.

This multi-morbidity is associated with polypharmacy, which is a recognised risk factor for poor treatment compliance.

One of the causes of poor compliance is a lack of understanding of the treatment. In this context, the role of the general practitioner is central. General practitioners are responsible for more than three-quarters of medical prescriptions. They are the ones who initiate first-line treatments for chronic diseases, but also the ones who renew treatments introduced by specialists.

DETAILED DESCRIPTION:
Objectives Primary: To describe the understanding of chronic treatments by patients over 65 years of age.

Secondary: To investigate the factors associated with the understanding of chronic treatments by patients over 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 65 or over
* Consulting one of the general practitioners agreeing to participate in the study
* Have a prescription containing at least one chronic treatment (defined as a treatment lasting more than 3 months)
* Agree to participate in the study.

Exclusion Criteria:

* Does not understand French,
* Has neurocognitive disorders
* Lives in a medical facility
* Consulting for an acute condition and whose prescription does not include chronic treatment.
* Protected by law (guardianship, curatorship, judicial protection),

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged over 65, not living in a care home, with a prescription containing at least one medicine prescribed as part of their chronic treatment, defined as lasting more than 3 months, and agreeing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Understanding each chronic treatment listed on the prescription | Day 0
  A complete understanding of each chronic treatment, defined by knowledge of the dosage (number of doses and timing) and the indication for chronic treatment

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Gestonnairedu CURRS, Reims, Université de Reims Champagne-Ardenne
  - Ufr Medecine Urca, Reims

IPD SHARING:
Plan to Share IPD: Undecided